CLINICAL TRIAL: NCT05664724
Title: Simultaneous Physiotherapy and Orthopedic Surgeon Interdisciplinary Care
Brief Title: Simultaneous Physiotherapy and Orthopedic Surgeon Interdisciplinary Care (SPOSIC)
Acronym: SPOSIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Interior Health (Industry)
Responsible Party: Principal Investigator, Brodie Sakakibara, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOSIC
Record Dates: First submitted 2022-12-01; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee; Arthritis
Keywords: arthroplasty; rehabilitation; interdisciplinary
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receives interdisciplinary sessions (Experimental): Interdisciplinary care by a team that includes: orthopedic surgeon, physiotherapist, a patient navigator, and the patient
  Interventions: Behavioral: Receives interdisciplinary sessions

INTERVENTIONS:
Behavioral: Receives interdisciplinary sessions — Along with usual care, participants receive six interdisciplinary sessions at 2 months and 1 month pre-operatively and 2 weeks, 6 weeks, 3 months, and 6 months post-operatively attended by an orthopedic surgeon, a physiotherapist, a patient navigator, and the patient. The pre-operative interdisciplinary sessions will outline expectations, explore patients' questions and concerns, set expectations for the next interdisciplinary session, and ensure goal congruence between all members of the team.
  Along with usual care during the post-operative period, participants will receive interdisciplinary sessions that address safety and medical issues, revisit patient expectations, reinforce care team expectations, focus on a personalized rehabilitation plan, and ensure goal congruence between the various team members.

SUMMARY:
This study will test a protocol to implement simultaneous physiotherapy and orthopedic surgeon interdisciplinary care for patients undergoing knee replacement surgery. These interdisciplinary sessions will help tailor personalized goals, involving the patient as a key member of the team.

DETAILED DESCRIPTION:
The purpose of this project is to test a quality improvement protocol to improve outcomes following knee arthroplasty surgery utilizing simultaneous physiotherapy and orthopedic surgeon interdisciplinary care. In an era of increasing demands on health care budgets, it is vital to improve quality of care without substantially increasing its cost. This study will focus on a quality improvement strategy that aims to redeploy existing resources to achieve higher quality care without substantially altering costs. This interdisciplinary approach involves establishing a high functioning team that includes the patient as a pivotal member and builds collaboration in the pre-operative period that can be leveraged in the post-operative period to achieve optimal outcomes. This differs from traditional, siloed care for knee arthroplasty.

Participants will be involved in usual care surrounding knee arthroplasty which includes education sessions and pre-habilitation pre-operatively and rehabilitation post-operatively. Participants will also attend two interdisciplinary sessions at 2 months and 1 month prior to surgery to outline expectations, explore patients' questions and concerns, set expectations for the next interdisciplinary session, and ensure goal congruence between all members of the team. At each of these sessions a physical assessment will also be completed by the orthopedic surgeon and physiotherapist. Following surgery, participants will attend four more interdisciplinary sessions at 2 weeks, 6 weeks, 3 months, and 6 months post-operatively. These sessions will address safety and medical issues, revisit patient expectations, reinforce care team expectations, focus on a personalized rehabilitation plan, and ensure goal congruence between the various team members. The physical assessment will also be repeated.

The objectives of the study are as follows:

1. Evaluate the feasibility (e.g., recruitment and retention, administrative and participant burden, lived experiences) of treating knee arthroplasty patients through a novel interdisciplinary program aimed to optimize recovery among patients; and
2. Estimate the size of the program's effect on biopsychosocial outcomes among community-dwelling individuals undergoing knee arthroplasty and rehabilitation.

The hypotheses of the study are as follows:

1. The protocol will establish proof-of-concept, and demonstrate sufficient feasibility to support a future full-scale multi-site RCT.
2. Simultaneous physiotherapy and orthopedic surgery interdisciplinary care (SPOSIC) will improve the primary outcome of functional disability, as measured by the 12-item Oxford Knee score (OKS), and improvements will also be shown in the secondary outcomes of pain, participation in social roles, health-related quality of life, and mobility.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. Expecting to undergo knee arthroplasty surgery within 12 months
3. Pain or functional limitation due to the musculoskeletal condition
4. Able to walk 10 meters without physical assistance
5. Able to tolerate 50 minutes of activity (including rest breaks, as needed)
6. Have adequate cognitive-communicative ability to participate (based on clinical judgment of the research team)
7. Able to provide informed consent

Exclusion Criteria:

1. Are living in long-term care
2. Have significant neurological conditions
3. Are medically unstable
4. Have medical condition(s) significantly impacting lower extremity function

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in Oxford Knee Score Questionnaire | Baseline, Post-intervention (immediately after 6 month post-op intervention)
  Subjectively measures functional ability. Minimum score: 0. Maximum score: 48. Higher score indicates better outcome.

SECONDARY OUTCOMES:
Change in Pain Visual Analogue Scale | Baseline, Post-intervention (immediately after 6 month post-op intervention)
  Subjective measurement of pain. Minimum score: 0cm. Maximum score: 10cm. Lower score indicates better outcome.
Change in Keele Assessment of Participation Questionnaire | Baseline, Post-intervention (immediately after 6 month post-op intervention)
  Subjective measurement of social role participation restrictions. Minimum score: 0. Maximum score: 44. Higher score indicates better outcome.
Change in EuroQol 5D3L Questionnaire | Baseline, Post-intervention (immediately after 6 month post-op intervention)
  Subjective measurement of health-related quality of life. Minimum score: 0.0. Maximum score: 1.0. Higher score indicates better outcome.
Change in Timed Up and Go Test | Baseline, Post-intervention (immediately after 6 month post-op intervention)
  Objectively measures mobility. Minimum score: 0s. Maximum score: unlimited s. A lower score indicates a better outcome.
Satisfaction Survey | Post-intervention (immediately after 6 month post-op intervention)
  Measures participants' satisfaction or dissatisfaction with the intervention. Scores ranked from strongly disagree to strongly agree. Strongly agree indicates a participant was more satisfied with the intervention.
Semi-structured interview | Post-intervention (immediately after 6 month post-op intervention)
  Open-ended questions regarding participants' attitudes and satisfaction with the program and areas for improvement

CONTACTS AND LOCATIONS:
Overall Officials: Brodie Sakakibara, PhD, Principal Investigator — The University of British Columbia

IPD SHARING:
Plan to Share IPD: No